CLINICAL TRIAL: NCT06512740
Title: The 2021-2022 Study of Family and Staff Well-Being in Head Start FACES Programs
Status: Completed | Type: Observational
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sara Bernstein, Principal Researcher, Mathematica Policy Research, Inc.
Other Study IDs: 51307-A
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Head Start Participation
Keywords: child care; child development; child health; child rearing; children; curriculum; early childhood education; families; Head Start; parenting; parents; parent well-being; teacher well-being; early childhood workforce; school readiness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head Start children and families: Children (1,837) Parents (1,837) Teachers (631) Program directors (176) Center directors (344)

SUMMARY:
The 2021-2022 Study of Family and Staff Well-Being in Head Start Family and Child Experiences Survey (FACES) Programs (the 2021-2022 Study) builds on FACES 2019, a national study of children and families participating in Head Start programs. In the year following the start of the COVID-19 pandemic, there was a need to understand how children, families, and Head Start staff were faring. The 2021-2022 Study explores child, family, and staff well-being, primarily in the programs that participated in FACES 2019.

DETAILED DESCRIPTION:
Since 1997, the Head Start Family and Child Experiences Survey (FACES) has been a source of information on the population in Head Start; staff qualifications, credentials, and opinions; Head Start classroom practices and characteristics; and the outcomes of children and families. The most recent nationally representative study was conducted in the 2019-2020 program year (entered as NCT03971435).

The motivation and goals of the Study of Family and Staff Well-Being in Head Start Family and Child Experiences Survey Programs (the 2021-2022 Study) came from a need that arose as the COVID-19 pandemic continued affecting Head Start families' and staff's lives into another program year. The Office of Planning, Research, and Evaluation in the Administration for Children and Families (ACF), U.S. Department of Health and Human Services, funded Mathematica and its partner-Juárez and Associates-to conduct a new data collection effort, the 2021-2022 Study, in fall and spring of the 2021-2022 Head Start program year. The goal was to provide data on the characteristics and needs of families and staff starting 18 months into the COVID-19 pandemic, and given heightened interest in the Head Start workforce.

The 2021-2022 Study includes data from a large multistage sample of Head Start programs, centers, teachers, and families from across the United States. Although the 2021-2022 Study selected a nationally representative sample of programs, centers, teachers, and children, fewer participated in the 2021-2022 Study than expected. Data from the 2021-2022 Study provide a window into the experiences of a sample of Head Start children, their families, and staff who were able to participate in data collection between October 2021 and July 2022. Readers should not assume the data are nationally representative of all Head Start programs, centers, teachers, families, or children. The data provide a snapshot of the experiences of Head Start staff, families, and children during this difficult time.

ELIGIBILITY:
The Head Start programs participating in the 2021-2022 Study were a probability sample selected from among 3,400 study-eligible programs on the 2017-2018 Head Start Program Information Report (PIR). To be eligible for the study, a program had to be:

* in one of the 50 states or the District of Columbia
* providing services directly to children ages 3 to 5 The Head Start Program Performance Standards require that children turn 3 by date used to determine eligibility for public school in the community in which the Head Start program is located. Therefore, some study children were 2 years old at the time of sampling if sampling occurred before the date used for public school eligibility.
* not be in imminent danger of losing its grantee status. Probability samples of centers were selected within each program, teachers within each center, and children within each teacher. Eligible teachers needed to have at least one Head Start child in their class.

Exclusion Criteria: American Indian and Alaska Native Head Start programs (Region XI) or Migrant and Seasonal Worker Head Start programs (Region XII) were not eligible.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Head Start children (and their families), Head Start programs, Head Start centers, Head Start classrooms/teachers.
Sampling Method: Probability Sample
Enrollment: 4825 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
General health status | October 2021-January 2022; April-July 2022
  Indicators of physical well-being were assessed by parent report to a survey item on if child's health is excellent, very good, good, fair, or poor
Social-emotional development | November 2021-January 2022; April-July 2022
  Indicators of social-emotional development were assessed using teacher report of several items on children's positive and problem behaviors. Please see the 2021-2022 Study User's Manual (Reid et al. 2024) for more information on the scores and technical information.
Social-emotional development - Approaches to learning | October 2021-January 2022; April-July 2022
  Indicators of social-emotional development were assessed using teacher and parent report of approaches to learning using the Early Childhood Longitudinal Study - Kindergarten Class of 1998 (ECLS-K). The items assess a child's motivation, attention, organization, persistence, and independence in learning. Please see U.S. Department of Education 2002 for more information on the scores and technical properties.
Parents' depressive symptoms | October 2021-January 2022; April-July 2022
  Parents' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Teachers' depressive symptoms | November 2021-January 2022; April-July 2022
  Teachers' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Program directors' depressive symptoms | April-July 2022
  Program directors' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Center directors' depressive symptoms | April-July 2022
  Center directors' levels of depressive symptoms were measured using the short form of the Center for Epidemiologic Studies-Depression Scale (CES-D). Please see Radloff 1977 for more information.
Parents' anxiety | October 2021-January 2022; April-July 2022
  Parents' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Teachers' anxiety | November 2021-January 2022; April-July 2022
  Teachers' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Program directors' anxiety | April-July 2022
  Program directors' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Center directors' anxiety | April-July 2022
  Center directors' anxiety levels were measured using items from the General Anxiety Disorder-7 (GAD-7). Please see Spitzer et al. 2006 for more information.
Staffing challenges | April-July 2022
  Staffing challenges were measured by summarizing center director survey items about the extent to which staff turnover has been a problem in terms of maintaining consistency in operations and care of children, and about finding classroom coverage and having enough staff to operate at full capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bernstein, Ph.D., Study Director — Mathematica Policy Research, Inc.; Nikki Aikens, Ph.D., Principal Investigator — Mathematica Policy Research, Inc.; Louisa Tarullo, Ed.D., Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Mathematica, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
In the future, he 2021-2022 Study of Family and Staff Well-Being in Head Start FACES Programs archived data will be available for access.
Time Frame: Data will become available within 2 years of completion.
Access Criteria: Applications for access to restricted-use data file include completing and adhering to a User Agreement.

REFERENCES:
- [Background] Radloff, L. "The CES-D Scale: A Self-Report Depression Scale for Research in the General Population." Applied Psychological Measurement, vol. 1, no. 3, 1977, pp. 385-401.
- [Background] Reid, M., A. Kopack Klein, E. Doran, B. Lepidus Carlson, J. Cannon, N. Aikens, S. Skidmore, K. Gonzalez, X. Li, L. Malone, S. Bernstein. "2021-2022 Study of Family and Staff Well-Being in Head Start FACES Programs (2021-2022 Study): User's Manual." Washington, DC: Mathematica, 2024.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] U.S. Department of Education, National Center for Education Statistics. Early Childhood Longitudinal Study-Kindergarten Class of 1998-99 (ECLS-K), Psychometric Report for Kindergarten through First Grade. NCES 2002-05. Washington, DC: National Center for Education Statistics, Institute of Education Sciences, U.S. Department of Education, 2002.